CLINICAL TRIAL: NCT03889015
Title: Comparison of Antibacterial Effect of Probiotic Yogurt Against Xylitol-containing Chewing Gum on Salivary Streptococcus Mutans Count, Bacterial Adherence and Salivary pH in Geriatric Patients: A Randomized Controlled Trial
Brief Title: Antibacterial Effect of Probiotic Yogurt Compared to Xylitol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadier Mahmoud Ahmed Gad, Internal resident in conservative department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: probiotic versus xylitol
Record Dates: First submitted 2019-03-16; First posted 2019-03-25 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Geriatric Patients

STUDY DESIGN:
Intervention Model Description: The subjects will be assigned randomly into two equal groups to receive either probiotic yogurt or xylitol-containing chewing gum for three months
Who Masked: Investigator, Outcomes Assessor
Masking Description: 1. Allocation concealment: Operator H.M. will choose between numbers in an opaque sealed envelope, which will be arranged by D.K. who will not be involved in any of the phases of the clinical trial. Data will be recorded on a computer by H.M. and O.S. and all records of all patients will be kept with the main supervisor M.I.
  2. Implementation: D.K. will generate the allocation sequence, enroll participants, and assign participants to interventions.
  3. Blinding: The assessors M.A. and R.E. will be blinded to the material assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- xylitol chewing gum (Active Comparator): Xylitol is widely used as an added sweetener in sugar-free products. It has been found to prevent dental caries through reducing dental plaque and limiting salivary streptococcus mutans counts and their produced levels of lactic acid
  Interventions: Dietary Supplement: xylitol chewing gum
- probiotic yogurt (Experimental): Probiotics are live microorganisms that confer oral health benefits by adhering to the oral mucosa and surface of teeth as a part of the biofilm thus preventing the adhesion, colonization, and proliferation of cariogenic bacteria inhibiting the formation of pathogenic plaque
  Interventions: Dietary Supplement: Probiotic yogurt

INTERVENTIONS:
Dietary Supplement: Probiotic yogurt — Probiotics are found in different dairy products including yoghurt, that are known as carriers of probiotics. These products can be easily integrated in daily meals to reduce cariogenic streptococcus mutans bacteria in dental biofilm
  Arms: probiotic yogurt
Dietary Supplement: xylitol chewing gum — Xylitol is widely used as an added sweetener in sugar-free products. It has been found to prevent dental caries through reducing dental plaque and limiting salivary streptococcus mutans counts and their produced levels of lactic acid
  Arms: xylitol chewing gum

SUMMARY:
This study will be conducted to evaluate the antibacterial effect of probiotic bacteria in yogurt in decreasing streptococcus mutans count in saliva and plaque, decreasing bacterial adherence and increasing salivary pH compared to xylitol-containing chewing gum after three months.

DETAILED DESCRIPTION:
The subjects will be assigned randomly into two equal groups to receive either probiotic yogurt or xylitol-containing chewing gum for three months. The probiotic yogurt is (Activia; Danone, Egypt) containing Bifidobacterium (7x107 CFU/g). The subjects assigned to probiotic yogurt group will be instructed to eat 100 g of the provided yogurt 10 minutes after dinner and not to brush their teeth until one hour later. The subjects assigned to the xylitol-chewing gum group will be instructed to chew the provided gum three times daily for five minutes after each meal.

ELIGIBILITY:
Inclusion Criteria:

* Above 50 years old.
* Have sufficient cognitive ability to understand consent procedures.
* Males or Females.
* Co-operative patients.
* High caries risk patients (≥105 CFU for streptococcus mutans count)

Exclusion Criteria:

* Under antibiotic treatment
* Milk intolerant
* Consuming any other probiotic product
* Habitual consumers of xylitol products
* Use antibacterial mouthwash
* Lack of compliance
* Any systemic condition affecting salivary secretion

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
streptococcus mutans count in saliva | 3 months
  The samples will be transported to the laboratory and cultured on selective media (dry Mitis Salivarius Agar with potassium tellurite medium and bacitracin) after serial dilutions. The plates will be incubated at 37ºC in 5-10% CO2 jar. then number of Colony Forming Units (CFU/ml) of Mutans Streptococci in saliva will be determined

SECONDARY OUTCOMES:
streptococcus mutans count in plaque | 3 months
  The samples will then be dispersed and spread over the culture media plates (mitis salivarius-bacitracin Agar), and the plates will be incubated under aerobic conditions
salivary pH | 3 months
  All the saliva samples will be tested on the same day for salivary pH using digital pH meter. The equipment will be calibrated with distilled water to reach pH 7 every time before measuring each sample
bacterial adherence | 3 months
  After applying disclosing agent over teeth, standard photographic images of the maxillary and mandibular facial surfaces of teeth will be taken. Digital plaque image analysis will be used to analyze plaque coverage. Images will be converted into pixels to calculate the percentage of the tooth covered with plaque divided by the total tooth area (both tooth areas with and without plaque) as follows:
  plaque area coverage = [plaque pixels / (tooth pixels + plaque pixels)] × 100 The computer analysis results will be checked for consistency and accuracy by an expert in image analysis who is blinded to the assigned treatment

IPD SHARING:
Plan to Share IPD: Undecided